CLINICAL TRIAL: NCT04061707
Title: Subcutaneous EEG: Forecasting of Epileptic Seizures Through Investigation of Long-term Dynamics of Seizure Occurrences, Stress, Sleep and Other Factors
Brief Title: Subcutaneous EEG: Forecasting of Epileptic Seizures
Acronym: SUBER
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS: 252686
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Epilepsies, Focal
Keywords: Focal Epilepsy; Longterm EEG Monitoring; Wearable Devices; mHealth; Seizure Forecasting
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Protocol Summary

Population - Target population is 10 adults (18 to 75 years of age) with a diagnosis of treatment-resistant epilepsy with at least 20 seizures per year, and whose seizure onset recorded from scalp EEG is localized to a brain region accessible by the subcutaneous EEG electrodes

Number of sites - Three sites; King's College Hospital NHS Foundation Trust, University College London Hospital NHS Foundation Trust, St George's University Hospital NHS Foundation Trust

Study design - This study is an observational, non-randomised, non-interventional study. It is not intended as a device trial. It is not intended to assess the device performance, rather the usefulness of bio-signals in seizure prediction and in detecting seizure-associated phenomena. There will be no change to usual care as a result of taking part.

A subcutaneous EEG device will be implanted under local anaesthesia to record continuous EEG and a non-invasive wrist-worn sensor will be used to acquire non-EEG bio-signals (eg. heart activity and rate, movements, muscle activity, electrodermal activity, body temperature)

Objectives - The association will be investigated between non-invasive measurable variables related to stress and sleep, semi-invasive subcutaneous EEG phenomena, and the occurrence of seizures. The predictive value of change in non-invasive variables semi-invasive subcutaneous EEG phenomena for the occurrence of seizures will be assessed.

Study Duration - Up to one year for each patient. Participants may be approached during or after this study to participate in related studies.

Funding - This study receives funding from the Epilepsy Foundation of America, Innovative Medicines Institute (IMI) and UNEEG medical A/S.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of treatment-resistant epilepsy of any syndrome, in which seizures are detectable in scalp EEG with two electrodes
* Between the ages of 18 - 75
* Experiencing >20 seizures (with impaired awareness) per year according to seizure diary.

Exclusion Criteria:

* Established current diagnosis of psychogenic non-epileptic attacks (dissociative seizures)
* Frequent vigorous involuntary movements (eg. chorea, athetosis) or frequent parasomnias with major motor components (eg. sleep walking, night terrors)
* Inability to comply with the trial procedure, such as cognitive or behavioral problems
* Inability to give informed consent
* History or evidence of: Severe cardiac disease (including Pacemaker and ICD-unit), Myocardial infarction, angina pectoris or other ischaemic heart disease, Cardiac arrhythmia or Any other heart failure
* History or evidence of: Stroke, Transient ischaemic attack, Carotid or vertebral artery stenosis or dissection, Cerebral hemorrhage, Any other structural cerebral disease
* Use of following drugs: Chemotherapeutic drugs of any kind, Methotrexate, Anticoagulation treatment, Immunosuppressant treatment, Third generation antipsychotic drugs (aripiprazole, quetiapine, clozapine, ziprasidone, paliperidone, risperidone, sertindole, amisulpride, olanzapine)
* Subjects under investigation or treatment of active cancer or cancer diagnosis within the past 5 years
* Subjects known with or suspected abuse of alcohol (defined as consumption of > 250g alcohol per week or abuse of any other neuro-active substances
* Subjects involved in therapies with medical devices that deliver electrical energy into the area around the implant.
* Subjects at high risk of surgical complications, such as active systemic infection and hemorrhagic disease.
* Subjects who are allergic to the local anesthetics used during implantation.
* Subjects whose safety blood measurements (full blood count, U&E, clotting) are significantly out of range in the judgement of the CI.
* Females of childbearing potential who are pregnant or intend to become pregnant or are not using adequate contraceptive methods throughout the study (Safe anticontraceptive methods includes contraceptive pills, intrauterine device including hormone intrauterine device and sustained gestagen injection)
* Subjects who have an infection at the site of device implantation.
* Subjects who operate MRI scanners or are planned to have an MRI scan within the next year.
* Subjects with profession/hobby that includes activity imposing extreme pressure variations (e.g. diving or parachute jumping). NB: diving/snorkeling is allowed to 5 meters of depth.
* Subjects with profession/hobby that includes activity imposing an unacceptable risk for trauma against the device or the site of implantation (e.g. martial art or boxing).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 10 suitable people with epilepsy referred, as part of their routine conventional care, to the Epilepsy Clinics at King's College Hospital (KCH), University College London Hospital NHS Foundation Trust (National Hospital for Neurology and Neurosurgery - NHNN), or St George's University Hospital NHS Foundation Trust (SGH).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Seizure Occurence | 1 year
  Proof-of-principle seizure-predictor based on continuously-acquired ultra-longterm subcutaneous EEG and non-invasive wearable sensor data

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Richardson, BM FRCP PhD, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No